CLINICAL TRIAL: NCT00976170
Title: A Phase I, Open-Label, Multi-center, Dose-escalation Study of the Safety, Tolerability, and Pharmacokinetics of GC33 in Combination With Sorafenib (Nexavar®) in Patients With Advanced or Metastatic Hepatocellular Carcinoma (HCC).
Brief Title: Study of GC33 and Sorafenib in Combination in Advanced or Metastatic Liver Cancer (Hepatocellular Carcinoma)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-002US
Record Dates: First submitted 2009-09-09; First posted 2009-09-14 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Advanced or metastatic HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — codrituzumab; Sorafenib

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: GC33(RO5137382); Drug: Sorafenib

INTERVENTIONS:
Drug: GC33(RO5137382) — IV administration at 6 escalating dose levels.
Drug: Sorafenib — Oral administration at 400mg twice daily or 400mg once daily

SUMMARY:
This phase I trial is studying the safety and best dose of GC33 and Sorafenib in combination in patients with advanced or metastatic liver cancer.

DETAILED DESCRIPTION:
This is a Phase I open-label dose escalation study of GC33 in combination with Sorafenib in patients with advanced or metastatic HCC. This study is designed to evaluate safety, tolerability, pharmacokinetics, and efficacy. Enrollment will proceed until a maximum tolerated dose (MTD) and a recommended Phase II dose has been established.

ELIGIBILITY:
Inclusion Criteria:

* Signed written Institutional Review Board/Ethical Committee approved informed consent form.
* Male or female ≥18 years old.
* Life expectancy ≥3 months.
* ECOG Performance Status of 0-1.
* Histologically confirmed hepatocellular carcinoma.
* Not a candidate for curative treatments.
* Child-Pugh A
* Hematological, Biochemical and Organ Function:

  * AST (SGOT): ≤5.0 × ULN,
  * ALT (SGPT): ≤5.0 × ULN,
  * Total Bilirubin: ≤1.5mg/dL,
  * Platelets: ≥100,000/μL,
  * Absolute Neutrophil Count: ≥1,500/μL,
  * Serum creatinine: ≤2.0 × ULN,
  * PT-INR: ≤2.0
* Ability to provide a tumor tissue sample either by:

  * A formalin fixed paraffin embedded block sample within 12 months prior to informed consent for HCC diagnosis
  * Undergo a biopsy to confirm HCC diagnosis
* Measurable disease.

Exclusion Criteria:

* Child-Pugh B or C
* Patient who have taken Sorafenib previously.
* Difficulty or inability to swallow pills.
* Pregnant or lactating women or women of child-bearing potential and men of childbearing potential not willing to use effective means of contraception.
* Patients known to be positive for Human immunodeficiency virus infection.
* Active infectious diseases requiring treatment except for hepatitis B and C.
* Other malignancies within the last 5 years.
* History of transplantation (organ, bone marrow transplantation, Peripheral blood stem cell transplantation, etc.).
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements..
* Patients with known brain metastases or other central nervous system disease/disorders.
* Uncontrolled hypertension defined as systolic blood pressure >150 mmhg or diastolic blood pressure >90 mmHg, despite optimal medical management.
* Non-tumor related thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Pulmonary hemorrhage/bleeding event ≥ CTCAE Grade 3, any other hemorrhage/bleeding event ≥ CTCAE Grade 4 within 4 weeks of first dose of study drug.
* Serious non-healing wound, ulcer, or bone fracture.
* Patients who received major surgery, local therapy for HCC, chemotherapy, radiotherapy, hormone-therapy, immunotherapy, or another investigational drug within 4 weeks prior to Day 1(6 weeks for nitrosoureas, mitomycin, and bevacizumab; 1 week for tumor biopsy).
* Patients who received the following treatments within 2 weeks prior to Day 1:

  * Anticoagulant or thrombolytic agents for therapeutic purposes,
  * Systemic anti-viral therapy for hepatitis C and Interferon therapy for hepatitis B,
  * Blood transfusion including all blood products
* Known history of hypersensitivity to similar agents.
* Patients receiving any medications or substances that are inducers of CYP3A4 are ineligible: rifampin, St. John's wort, phenytoin, carbamazepine, phenobarbital and dexamethasone.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol requirements and/or follow-up procedures; those conditions should be discussed with the patient before trial entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2013-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Toxicity evaluation in accordance with CTCAE v3.0 | Continuous
Dose limiting toxicity and maximum tolerated dose | Continuous

SECONDARY OUTCOMES:
RECIST criteria (version 1.0) for response evaluation by CT/MRI in target and non-target lesions of HCC | every 2 months
Repeat-dose pharmacokinetic behavior of GC33 and Sorafenib | Continuous

CONTACTS AND LOCATIONS:
Locations (7):
- United States (5):
  - California Pacific Medical Center, San Francisco, California
  - University of Miami, Miami, Florida
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan Univercity Hospital, Taipei

REFERENCES:
- [Derived] Abou-Alfa GK, Yen CJ, Hsu CH, O'Donoghue J, Beylergil V, Ruan S, Pandit-Taskar N, Gansukh B, Lyashchenko SK, Ma J, Wan P, Shao YY, Lin ZZ, Frenette C, O'Neil B, Schwartz L, Smith-Jones PM, Ohtomo T, Tanaka T, Morikawa H, Maki Y, Ohishi N, Chen YC, Agajanov T, Boisserie F, Di Laurenzio L, Lee R, Larson SM, Cheng AL, Carrasquilo JA. Phase Ib study of codrituzumab in combination with sorafenib in patients with non-curable advanced hepatocellular carcinoma (HCC). Cancer Chemother Pharmacol. 2017 Feb;79(2):421-429. doi: 10.1007/s00280-017-3241-9. Epub 2017 Jan 24. PMID 28120036